CLINICAL TRIAL: NCT02445937
Title: Stepped Wedge Trial of an Intervention to Support Proxy Decision Makers in ICUs
Brief Title: PARTNER II: Improving Patient and Family Centered Care in Advanced Critical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Douglas White, Vice Chair and Professor of Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO14090204
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Anxiety; Depression
Keywords: decision making for incapacitated patients; intensive care; surrogate decision making; patient centered care; palliative care
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): The control group will receive usual care, in which the frequency and content of physician-family communication is determined by the clinical team according to their usual practice. No study ICU has a protocolized approach to family communication and instead clinicians determine the timing and frequency of communication with families. All sites have palliative care services.
- Behavioral: The PARTNER II Intervention (Experimental): The PARTNER intervention is a multifaceted intervention delivered by a trained "PARTNER Champion" who has undergone 16 hours of intense communication training, with audit and feedback, quarterly booster training, and expert implementation support. Additionally, there is academic detailing of ICU physicians and ICU bedside nurses to augment the intervention. The PARTNER Intervention deploys three strategies to improve: 1) the timeliness and frequency of clinician-family communication, 2) the emotional and decision support provided to families and 3) the appropriate involvement of palliative care specialists.
  Interventions: Behavioral: PARTNER II

INTERVENTIONS:
Behavioral: PARTNER II — The PARTNER intervention is a multifaceted intervention delivered by a trained "PARTNER Champion" who has undergone 16 hours of intense communication training, with audit and feedback, quarterly booster training, and expert implementation support. Additionally, there is academic detailing of ICU physicians and ICU bedside nurses to augment the intervention. The PARTNER Intervention deploys three strategies to improve: 1) the timeliness and frequency of clinician-family communication, 2) the emotional and decision support provided to families and 3) the appropriate involvement of palliative care specialists.
  Arms: Behavioral: The PARTNER II Intervention

SUMMARY:
This is a stepped wedged randomized controlled trial comparing the PARTNER intervention with usual care in 5 Intensive Care Units. The overarching goal of this research project to ensure patient-centered decisions about the use of intensive treatments for patients with advanced critical illness. In a prior project, the investigators developed the PARTNER program (PAiring Re-engineered ICU Teams with Nurse-driven Education and OutReach), a 4-facet, team-based intervention that re-engineers how surrogates are supported in ICUs, including: 1) changing care "defaults" to ensure clinician-family meetings within 48 hours of enrollment and frequently thereafter; 2) protocolized, nurse-administered coaching and emotional support of surrogates before and during clinician-family meetings, 3) increased use of palliative care services for patients with a poor prognosis. The investigators propose to begin deployment of the PARTNER II program in the spring of 2015 enrolling 690 surrogate decision makers in 5 ICUs using a stepped wedge design. The investigators expect to achieve the following project goals:

1. To increase the patient-centeredness of end-of-life decisions, and to increase the quality of clinician-family communication.
2. To decrease the psychological burden on family members acting as surrogates.
3. To reduce total health care costs by decreasing the duration of use of burdensome, invasive treatments at the end of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Surrogate decision maker for ICU patient in one of 5 UPMC ICU's

Exclusion Criteria:

* Non-English Speaking
* Surrogate's loved one is for organ transplantation
* Not physically able to participate in family meeting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Quality of Communication (QOC) scale | At 6 months
  We will assess quality of communication in family members in a telephone interview 6 months after enrollment using the validated13 item Quality of Communication Scale.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | At 6 months
  We will assess symptom burden of anxiety and depression in family members in a telephone interview 6 months after enrollment using the validated 14-item Hospital Anxiety and Depression scale (HADS).
Patient-Centeredness of Care Scale | At 6 months
  We will assess Patient Centeredness of Care, using the 12-item Patient-Perceived Patient-Centeredness of Care Scale (PPPC) adapted for use by surrogates.
Intensive Care Unit Length of Stay | Participants will be followed for duration of ICU stay, an expected average of 21 days
  We will assess the Intensive Care Unit length of stay as assessed by abstraction of this information from the medical record.
Impact of Events Scale | At 6 months
  We will assess symptoms of post-traumatic stress in family members in a telephone interview 6 months after enrollment using the validated 22 item Impact of Events Scale.
Decision Regret Scale | At 6 months
  We will assess Decisional Regret by family members in a telephone interview 6 months after enrollment using the validated 5 item Decision Regret Scale across treatment groups.

OTHER OUTCOMES:
Mortality | At 6 months
  We will assess hospital mortality and 6-month mortality using hospital records, 6 month follow-up with surrogates, and the National Death Index in cases in which participants are lost to telephone follow up.
Katz Activities of Daily Living Scale | At 6 months
  We will assess functional status of the patient using the validated Katz Activities of Daily Living Scale at 6 months.
Hospital Length of Stay | Participants will be followed for duration of hospital stay, an expected average of 4 weeks.
  We will assess hospital length of stay by abstraction of this information from the medical record at hospital discharge.
Total Hospitalization costs | Inclusive of index hospitalization
  We will measure total hospitalization costs by aggregating each patient's total service specific costs, generated from hospital administrative records.
6-month health care utilization | Inclusive of index hospitalization and 6 months follow up
  We will assess patient health care utilization using hospital records and through validated methods to assess utilization using standardized interviews with surrogates at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B. White, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Hamot, Erie, Pennsylvania
  - UPMC Presby/Shady, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Angus DC, Barnato AE, Linde-Zwirble WT, Weissfeld LA, Watson RS, Rickert T, Rubenfeld GD; Robert Wood Johnson Foundation ICU End-Of-Life Peer Group. Use of intensive care at the end of life in the United States: an epidemiologic study. Crit Care Med. 2004 Mar;32(3):638-43. doi: 10.1097/01.ccm.0000114816.62331.08. PMID 15090940
- [Background] Prendergast TJ, Claessens MT, Luce JM. A national survey of end-of-life care for critically ill patients. Am J Respir Crit Care Med. 1998 Oct;158(4):1163-7. doi: 10.1164/ajrccm.158.4.9801108. PMID 9769276
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Wendler D, Rid A. Systematic review: the effect on surrogates of making treatment decisions for others. Ann Intern Med. 2011 Mar 1;154(5):336-46. doi: 10.7326/0003-4819-154-5-201103010-00008. PMID 21357911
- [Background] Lynn J, Teno JM, Phillips RS, Wu AW, Desbiens N, Harrold J, Claessens MT, Wenger N, Kreling B, Connors AF Jr. Perceptions by family members of the dying experience of older and seriously ill patients. SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. Ann Intern Med. 1997 Jan 15;126(2):97-106. doi: 10.7326/0003-4819-126-2-199701150-00001. PMID 9005760
- [Background] Murphy DJ, Burrows D, Santilli S, Kemp AW, Tenner S, Kreling B, Teno J. The influence of the probability of survival on patients' preferences regarding cardiopulmonary resuscitation. N Engl J Med. 1994 Feb 24;330(8):545-9. doi: 10.1056/NEJM199402243300807. PMID 8302322
- [Background] Weeks JC, Cook EF, O'Day SJ, Peterson LM, Wenger N, Reding D, Harrell FE, Kussin P, Dawson NV, Connors AF Jr, Lynn J, Phillips RS. Relationship between cancer patients' predictions of prognosis and their treatment preferences. JAMA. 1998 Jun 3;279(21):1709-14. doi: 10.1001/jama.279.21.1709. PMID 9624023
- [Background] Riley GF, Lubitz JD. Long-term trends in Medicare payments in the last year of life. Health Serv Res. 2010 Apr;45(2):565-76. doi: 10.1111/j.1475-6773.2010.01082.x. Epub 2010 Feb 9. PMID 20148984
- [Background] Hogan C, Lunney J, Gabel J, Lynn J. Medicare beneficiaries' costs of care in the last year of life. Health Aff (Millwood). 2001 Jul-Aug;20(4):188-95. doi: 10.1377/hlthaff.20.4.188. PMID 11463076
- [Background] Fried TR, Bradley EH, Towle VR, Allore H. Understanding the treatment preferences of seriously ill patients. N Engl J Med. 2002 Apr 4;346(14):1061-6. doi: 10.1056/NEJMsa012528. PMID 11932474
- [Background] Sudore RL, Fried TR. Redefining the "planning" in advance care planning: preparing for end-of-life decision making. Ann Intern Med. 2010 Aug 17;153(4):256-61. doi: 10.7326/0003-4819-153-4-201008170-00008. PMID 20713793
- [Background] Schneiderman LJ, Gilmer T, Teetzel HD, Dugan DO, Blustein J, Cranford R, Briggs KB, Komatsu GI, Goodman-Crews P, Cohn F, Young EW. Effect of ethics consultations on nonbeneficial life-sustaining treatments in the intensive care setting: a randomized controlled trial. JAMA. 2003 Sep 3;290(9):1166-72. doi: 10.1001/jama.290.9.1166. PMID 12952998
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Background] Bedell SE, Pelle D, Maher PL, Cleary PD. Do-not-resuscitate orders for critically ill patients in the hospital. How are they used and what is their impact? JAMA. 1986 Jul 11;256(2):233-7. PMID 3723709
- [Background] Eidelman LA, Jakobson DJ, Pizov R, Geber D, Leibovitz L, Sprung CL. Foregoing life-sustaining treatment in an Israeli ICU. Intensive Care Med. 1998 Feb;24(2):162-6. doi: 10.1007/s001340050539. PMID 9539075
- [Background] Faber-Langendoen K. The clinical management of dying patients receiving mechanical ventilation. A survey of physician practice. Chest. 1994 Sep;106(3):880-8. doi: 10.1378/chest.106.3.880. PMID 8082372
- [Background] Keenan SP, Busche KD, Chen LM, McCarthy L, Inman KJ, Sibbald WJ. A retrospective review of a large cohort of patients undergoing the process of withholding or withdrawal of life support. Crit Care Med. 1997 Aug;25(8):1324-31. doi: 10.1097/00003246-199708000-00019. PMID 9267945
- [Background] Koch KA, Rodeffer HD, Wears RL. Changing patterns of terminal care management in an intensive care unit. Crit Care Med. 1994 Feb;22(2):233-43. doi: 10.1097/00003246-199402000-00013. PMID 8306681
- [Background] Smedira NG, Evans BH, Grais LS, Cohen NH, Lo B, Cooke M, Schecter WP, Fink C, Epstein-Jaffe E, May C, et al. Withholding and withdrawal of life support from the critically ill. N Engl J Med. 1990 Feb 1;322(5):309-15. doi: 10.1056/NEJM199002013220506. PMID 2296273
- [Background] Vernon DD, Dean JM, Timmons OD, Banner W Jr, Allen-Webb EM. Modes of death in the pediatric intensive care unit: withdrawal and limitation of supportive care. Crit Care Med. 1993 Nov;21(11):1798-802. doi: 10.1097/00003246-199311000-00035. PMID 7802736
- [Background] Vincent JL, Parquier JN, Preiser JC, Brimioulle S, Kahn RJ. Terminal events in the intensive care unit: review of 258 fatal cases in one year. Crit Care Med. 1989 Jun;17(6):530-3. doi: 10.1097/00003246-198906000-00009. PMID 2721211
- [Background] Youngner SJ, Lewandowski W, McClish DK, Juknialis BW, Coulton C, Bartlett ET. 'Do not resuscitate' orders. Incidence and implications in a medical-intensive care unit. JAMA. 1985 Jan 4;253(1):54-7. doi: 10.1001/jama.253.1.54. PMID 3964898
- [Background] Sprung CL, Cohen SL, Sjokvist P, Baras M, Bulow HH, Hovilehto S, Ledoux D, Lippert A, Maia P, Phelan D, Schobersberger W, Wennberg E, Woodcock T; Ethicus Study Group. End-of-life practices in European intensive care units: the Ethicus Study. JAMA. 2003 Aug 13;290(6):790-7. doi: 10.1001/jama.290.6.790. PMID 12915432
- [Background] Prendergast TJ, Luce JM. Increasing incidence of withholding and withdrawal of life support from the critically ill. Am J Respir Crit Care Med. 1997 Jan;155(1):15-20. doi: 10.1164/ajrccm.155.1.9001282.
- [Background] Kirchhoff KT, Walker L, Hutton A, Spuhler V, Cole BV, Clemmer T. The vortex: families' experiences with death in the intensive care unit. Am J Crit Care. 2002 May;11(3):200-9. PMID 12022483
- [Background] Tilden VP, Tolle SW, Garland MJ, Nelson CA. Decisions about life-sustaining treatment. Impact of physicians' behaviors on the family. Arch Intern Med. 1995 Mar 27;155(6):633-8. PMID 7887760
- [Background] Tilden VP, Tolle SW, Nelson CA, Fields J. Family decision-making to withdraw life-sustaining treatments from hospitalized patients. Nurs Res. 2001 Mar-Apr;50(2):105-15. doi: 10.1097/00006199-200103000-00006. PMID 11302290
- [Background] A controlled trial to improve care for seriously ill hospitalized patients. The study to understand prognoses and preferences for outcomes and risks of treatments (SUPPORT). The SUPPORT Principal Investigators. JAMA. 1995 Nov 22-29;274(20):1591-8. PMID 7474243
- [Background] Hofmann JC, Wenger NS, Davis RB, Teno J, Connors AF Jr, Desbiens N, Lynn J, Phillips RS. Patient preferences for communication with physicians about end-of-life decisions. SUPPORT Investigators. Study to Understand Prognoses and Preference for Outcomes and Risks of Treatment. Ann Intern Med. 1997 Jul 1;127(1):1-12. doi: 10.7326/0003-4819-127-1-199707010-00001. PMID 9214246
- [Background] Curtis JR, Engelberg RA, Bensink ME, Ramsey SD. End-of-life care in the intensive care unit: can we simultaneously increase quality and reduce costs? Am J Respir Crit Care Med. 2012 Oct 1;186(7):587-92. doi: 10.1164/rccm.201206-1020CP. Epub 2012 Aug 2. PMID 22859524
- [Background] Luce JM, Rubenfeld GD. Can health care costs be reduced by limiting intensive care at the end of life? Am J Respir Crit Care Med. 2002 Mar 15;165(6):750-4. doi: 10.1164/ajrccm.165.6.2109045. No abstract available. PMID 11897638
- [Background] White DB, Arnold RM. The evolution of advance directives. JAMA. 2011 Oct 5;306(13):1485-6. doi: 10.1001/jama.2011.1430. No abstract available. PMID 21972313
- [Background] Hawkins NA, Ditto PH, Danks JH, Smucker WD. Micromanaging death: process preferences, values, and goals in end-of-life medical decision making. Gerontologist. 2005 Feb;45(1):107-17. doi: 10.1093/geront/45.1.107. PMID 15695421
- [Background] Song MK, Ward SE, Happ MB, Piraino B, Donovan HS, Shields AM, Connolly MC. Randomized controlled trial of SPIRIT: an effective approach to preparing African-American dialysis patients and families for end of life. Res Nurs Health. 2009 Jun;32(3):260-73. doi: 10.1002/nur.20320. PMID 19205027
- [Background] Danis M. Improving end-of-life care in the intensive care unit: what's to be learned from outcomes research? New Horiz. 1998 Feb;6(1):110-8. PMID 9508265
- [Background] Institute of Medicine (US) Committee on Identifying Priority Areas for Quality Improvement; Adams K, Corrigan JM, editors. Priority Areas for National Action: Transforming Health Care Quality. Washington (DC): National Academies Press (US); 2003. Available from http://www.ncbi.nlm.nih.gov/books/NBK221294/ PMID 25057643
- [Background] Institute of Medicine (US) Committee on the Robert Wood Johnson Foundation Initiative on the Future of Nursing, at the Institute of Medicine. The Future of Nursing: Leading Change, Advancing Health. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209880/ PMID 24983041
- [Derived] Lincoln T, Shields AM, Buddadhumaruk P, Chang CH, Pike F, Chen H, Brown E, Kozar V, Pidro C, Kahn JM, Darby JM, Martin S, Angus DC, Arnold RM, White DB. Protocol for a randomised trial of an interprofessional team-delivered intervention to support surrogate decision-makers in ICUs. BMJ Open. 2020 Mar 29;10(3):e033521. doi: 10.1136/bmjopen-2019-033521. PMID 32229520